CLINICAL TRIAL: NCT05008939
Title: Subanesthetic Sevoflurane for Treatment-Resistant Depression: A Proof-of-Concept Trial
Brief Title: Sevoflurane for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: Shanghai Pudong New Area Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShanghaiFMIH2021 Zhiqiang Liu
Record Dates: First submitted 2021-07-25; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major
Keywords: treatment-resistant depression (TRD); major depressive disorder (MDD); sevoflurane
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Sevoflurane; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane (Experimental): Those with 1-hour inhalation of 1% sevoflurane/30% oxygen
  Interventions: Drug: Sevoflurane; Drug: Placebo
- placebo (Placebo Comparator): Those with 1-hour inhalation of 30% oxygen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sevoflurane — Patients receive 1% sevoflurane and 30% oxygen for 1 hour.
  Other Names: Treatment
  Arms: sevoflurane
Drug: Placebo — Patients received 30% oxygen for 1 hour.
  Other Names: Control

SUMMARY:
This study intends to carry out a prospective, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of subanesthetic sevoflurane for treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years
2. meeting DSM-V criteria for major depressive disorder
3. a pretreatment score ≥17 on HDRS-17
4. meeting criteria for TRD, defined as having had at least two adequate dose-duration antidepressant medication failures in the current depressive episode.
5. current treatment drugs were stably used for at least 4 weeks

Exclusion Criteria:

1. MDD with psychosis, e.g., bipolar disorder, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, panic disorder, et al
2. Drug, tobacco or alcohol abuse
3. active suicidal intention
4. previous administration of NMDA receptor antagonists (e.g., ketamine)
5. previous (<6 weeks prior) or ongoing treatment with electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS)
6. pregnancy or breastfeeding
7. morbidly obese, BMI>35kg/m2
8. other diseases that could interfere with the results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Rates of treatment responses in 17-item Hamilton Depression Rating Scale (HDRS-17) | 24 hours after the end of treatment
  ≥50% HDRS-17 reduction in depressive symptoms

SECONDARY OUTCOMES:
Rates of treatment responses in HDRS-17 | 2 hours, 7 days,14 days and 28 days after the end of treatment
  ≥50% HDRS-17 reduction in depressive symptoms
Rates of remissions in HDRS-17 | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  HDRS-17 ≤7 points
Rates of treatment responses in Montgomery-Åsberg Depression Rating Scale (MADRS) | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  ≥50% MADRS reduction in the baseline score
Rates of remissions in MADRS | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  MADRS <10
The assessment of depression with self-rating scale | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  The changes of score in Patient Health Questionnaire-9 (PHQ-9)
The assessment of anxiety by psychiatrist | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  The changes of score in Hamilton Anxiety Rating Scale (HAMA)
The assessment of anxiety with self-rating scale | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  The changes of score in Generalized Anxiety Disorder Screener (GAD-7)
The assessment of improvement by psychiatrist | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  The changes of score in Clinical Global Impression (CGI)
The assessment of improvement with self-rating scale | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  The changes of score in Patient Global Impressions of Improvement (PGI-I)
The assessment of side effects with self-rating scale | 2 hours, 24 hours, 7 days,14 days and 28 days after the end of treatment
  Including Patient Rated Inventory of Side Effects (PRISE)
Side effects of sevoflurane | up to 2 hours after the end of treatment
  Including nausea, vomiting, headache, dizzy, hypotension, hypoxemia, carbon dioxide accumulation, et al

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Liu, MD, Study Chair — Department of Anesthesiaology, Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaynes BN, Warden D, Trivedi MH, Wisniewski SR, Fava M, Rush AJ. What did STAR*D teach us? Results from a large-scale, practical, clinical trial for patients with depression. Psychiatr Serv. 2009 Nov;60(11):1439-45. doi: 10.1176/ps.2009.60.11.1439. PMID 19880458
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Background] Mrazek DA, Hornberger JC, Altar CA, Degtiar I. A review of the clinical, economic, and societal burden of treatment-resistant depression: 1996-2013. Psychiatr Serv. 2014 Aug 1;65(8):977-87. doi: 10.1176/appi.ps.201300059. PMID 24789696
- [Background] Papakostas GI, Petersen TJ, Farabaugh AH, Murakami JL, Pava JA, Alpert JE, Fava M, Nierenberg AA. Psychiatric comorbidity as a predictor of clinical response to nortriptyline in treatment-resistant major depressive disorder. J Clin Psychiatry. 2003 Nov;64(11):1357-61. doi: 10.4088/jcp.v64n1112. PMID 14658951
- [Background] Collins PY, Patel V, Joestl SS, March D, Insel TR, Daar AS; Scientific Advisory Board and the Executive Committee of the Grand Challenges on Global Mental Health; Anderson W, Dhansay MA, Phillips A, Shurin S, Walport M, Ewart W, Savill SJ, Bordin IA, Costello EJ, Durkin M, Fairburn C, Glass RI, Hall W, Huang Y, Hyman SE, Jamison K, Kaaya S, Kapur S, Kleinman A, Ogunniyi A, Otero-Ojeda A, Poo MM, Ravindranath V, Sahakian BJ, Saxena S, Singer PA, Stein DJ. Grand challenges in global mental health. Nature. 2011 Jul 6;475(7354):27-30. doi: 10.1038/475027a. No abstract available. PMID 21734685
- [Background] Berlim MT, Turecki G. Definition, assessment, and staging of treatment-resistant refractory major depression: a review of current concepts and methods. Can J Psychiatry. 2007 Jan;52(1):46-54. doi: 10.1177/070674370705200108. PMID 17444078
- [Background] Sanacora G, Schatzberg AF. Ketamine: promising path or false prophecy in the development of novel therapeutics for mood disorders? Neuropsychopharmacology. 2015 Mar 13;40(5):1307. doi: 10.1038/npp.2014.338. No abstract available. PMID 25767082
- [Background] Chen C, Ji M, Xu Q, Zhang Y, Sun Q, Liu J, Zhu S, Li W. Sevoflurane attenuates stress-enhanced fear learning by regulating hippocampal BDNF expression and Akt/GSK-3beta signaling pathway in a rat model of post-traumatic stress disorder. J Anesth. 2015 Aug;29(4):600-8. doi: 10.1007/s00540-014-1964-x. Epub 2014 Dec 23. PMID 25533726
- [Background] Zhang H, Li L, Sun Y, Zhang X, Zhang Y, Xu S, Zhao P, Liu T. Sevoflurane prevents stroke-induced depressive and anxiety behaviors by promoting cannabinoid receptor subtype I-dependent interaction between beta-arrestin 2 and extracellular signal-regulated kinases 1/2 in the rat hippocampus. J Neurochem. 2016 May;137(4):618-29. doi: 10.1111/jnc.13613. Epub 2016 Mar 31. PMID 26991409
- [Background] Luo C, Zhang YL, Luo W, Zhou FH, Li CQ, Xu JM, Dai RP. Differential effects of general anesthetics on anxiety-like behavior in formalin-induced pain: involvement of ERK activation in the anterior cingulate cortex. Psychopharmacology (Berl). 2015 Dec;232(24):4433-44. doi: 10.1007/s00213-015-4071-2. Epub 2015 Sep 24. PMID 26400403
- [Background] Guo Z, Zhao F, Wang Y, Wang Y, Geng M, Zhang Y, Ma Q, Xu X. Sevoflurane Exerts an Anti-depressive Action by Blocking the HMGB1/TLR4 Pathway in Unpredictable Chronic Mild Stress Rats. J Mol Neurosci. 2019 Dec;69(4):546-556. doi: 10.1007/s12031-019-01380-2. Epub 2019 Jul 31. PMID 31368063